CLINICAL TRIAL: NCT03622281
Title: Quality Improvement Intervention in Colonoscopy Using Artificial Intelligence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018SDU-QILU-716
Record Dates: First submitted 2018-07-16; First posted 2018-08-09 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Quality Control; Artificial Intelligence; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopists who received quality intervention (Experimental)
  Interventions: Other: quality improvement intervention using artificial intelligence
- Colonoscopists who did not received quality intervention (No Intervention)

INTERVENTIONS:
Other: quality improvement intervention using artificial intelligence — Colonoscopists received performance measure monitoring and feedback
  Arms: Colonoscopists who received quality intervention

SUMMARY:
Quality measures in colonoscopy are important guides for improving the quality of patient care. But quality improvement intervention is not taking place, primarily because of the inconvenience and expense. To address the difficulties above, we used artificial intelligence for quality control of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80;
* agree to give written informed consent.

Exclusion Criteria:

* patients with the contraindications to colonoscopy examination;
* patients with a history of inflammatory bowel disease (IBD), CRC, colorectal surgery;
* patients with prior failed colonoscopy and high suspicion of polyposis syndromes, IBD and typical advanced CRC;
* patients refused to participate in the trial;
* the colonoscopyprocedure cannot be completed due to stenosis, obstruction, huge occupying lesions, or solid stool;
* the colonoscopy procedure have to be terminated due to complications of anaesthesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 8 months
  Adenoma detection rate was defined as the number of exams with findings of adenoma divided by the total number of exams.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Su JR, Li Z, Shao XJ, Ji CR, Ji R, Zhou RC, Li GC, Liu GQ, He YS, Zuo XL, Li YQ. Impact of a real-time automatic quality control system on colorectal polyp and adenoma detection: a prospective randomized controlled study (with videos). Gastrointest Endosc. 2020 Feb;91(2):415-424.e4. doi: 10.1016/j.gie.2019.08.026. Epub 2019 Aug 24. PMID 31454493